CLINICAL TRIAL: NCT03625076
Title: Intra-articular Lidocaine vs Procedural Sedation for Anterior Shoulder Dislocations
Brief Title: IAL vs PS for Anterior Shoulder Dislocations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kendall Healthcare Group, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-233-Non-NSU Health
Record Dates: First submitted 2018-06-18; First posted 2018-08-10 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Lidocaine; Etomidate; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intra-articular Lidocaine (Experimental): 20 mL of 1% lidocaine injected into the joint of the dislocated shoulder
  Interventions: Drug: Intra-articular Lidocaine
- Procedural Sedation (Active Comparator): Intravenous etomidate or propofol
  Interventions: Drug: Procedural Sedation with etomidate or propofol

INTERVENTIONS:
Drug: Intra-articular Lidocaine — 20 mL of 1% Lidocaine will be injected into the joint of the dislocated shoulder. Afterwards, the physician will attempt to reduce the shoulder using a technique of his or her choice.
  Arms: Intra-articular Lidocaine
Drug: Procedural Sedation with etomidate or propofol — Procedural sedation using etomidate or propofol (physician's choice) will be performed. The dose of the drugs will also be left the treating physician. The physician will then attempt to reduce the shoulder using a technique of his or her choice.
  Arms: Procedural Sedation

SUMMARY:
This study compares intra-articular lidocaine to procedural sedation for the reduction of anterior shoulder dislocations in the emergency department.

DETAILED DESCRIPTION:
This will be a single center, prospective, open-label, randomized controlled trial on a convenience sample of patients presenting to the ED with anterior shoulder dislocations. This study will enroll all patients between the ages of 18 and 70 who meet all of the inclusion criteria and do not meet any of the exclusion criteria, who present to the ED with an anterior shoulder dislocation as determined by the ED physician. Written, informed consent will be obtained from each patient. After enrollment, each patient will be randomized either to IV sedation (with the provider's choice of propofol or etomidate) or intra-articular lidocaine. Randomization will be done before the initiation of data collection, and will be done with a random number generator. Patients who are randomized to the intra-articular group will receive 20 mL of 1% lidocaine injected into the glenohumeral joint using a lateral approach. Treating clinicians will be instructed to wait 10 minutes after injection before attempting reduction. The primary outcome measure will be the difference in emergency department length of stay between the procedural sedation and intra-articular lidocaine groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-70 years old in the emergency department with an anterior shoulder dislocation.

Exclusion Criteria:

* Pregnant or breastfeeding
* Is a prisoner.
* Known allergy to one of the study drugs.
* Altered mental status.
* Shoulder fracture (other than a Hill-Sachs) associated with the dislocation.
* Attending provider excludes patient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-05-02 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Emergency Department Length of Stay | Anticipated 1-4 hours
  The elapsed time over which the patient is physically in the emergency department

SECONDARY OUTCOMES:
Number of Reduction Attempts | Each attempt takes under 5 minutes
  The number of attempts it took the physician to reduce the shoulder dislocation
Patient Satisfaction | The patient is asked their satisfaction just prior to discharge (generally within 4 hours)
  The patient's satisfaction on a scale from 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Kendall Regional Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
If, after data collection, we feel that the release of IPD will increase the clarity of our data, we might make IPD available to other researchers.